CLINICAL TRIAL: NCT02825303
Title: Mid-term Effect of a Novel Sit-to-stand Workplace (ACTIVE OFFICE) on Cognitive and Physiological Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences Upper Austria (Other)
Collaborators: University of Vienna (Other)
Responsible Party: Principal Investigator, Bernhard Schwartz, Research Associate, University of Applied Sciences Upper Austria
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AO-8735-1; 834185 (Other Grant/Funding Number: Austrian Research Promotion Agency (FFG))
Record Dates: First submitted 2016-07-04; First posted 2016-07-07 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Sedentary Lifestyle; Worksite
Keywords: postural changes; Height adjustable desk; Prolonged sitting; Cognitive performance
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Novel workplace - first half (Experimental): Intervention: A novel two-desk sit-to-stand workstation for 23 weeks; provided within the first half of the study. Traditional workstation within the second half of the study.
  Interventions: Other: Workplace consisting of two height-adjustable desks
- Novel workplace - second half (Experimental): Intervention: A novel two-desk sit-to-stand workstation for 23 weeks; provided within the second half of the study. Traditional workstation within the frist half of the study.
  Interventions: Other: Workplace consisting of two height-adjustable desks
- Control group (No Intervention): Control group subjects did not encounter any changes in their regular office environments. Traditional workstation for both halves of the study.

INTERVENTIONS:
Other: Workplace consisting of two height-adjustable desks — Desk arrangements: self-determined by the participants Desk equipment: depending on pre-intervention condition - 1 or 2 screens per desk Build-up: one day prior to the intervention period at the location of the workplace Adjustment: together with the study leader
  Arms: Novel workplace - first half; Novel workplace - second half

SUMMARY:
Prolonged sitting is a risk factor for cardiovascular and musculoskeletal diseases, diabetes, several types of cancer and all-cause mortality. In combination with static and awkward postures, the prevalence of musculoskeletal diseases can increase further. Although the implementation of sit-to-stand or active workstations can help to reduce sitting time, improve physical activity at work and promote health benefits, it might also lead to changes in cognitive functions such as productivity The purpose of this study is to evaluate the mid-term effect of a novel two desk sit-to-stand workplace on sitting time as well as physiological and cognitive parameters for healthy people of working age in comparison to their traditional workplace.

DETAILED DESCRIPTION:
Measurements were made both in the field and in a laboratory. Field measurements were made and processed continuously over the 23-week intervention period. Laboratory measurements were made on two different days, one day prior to intervention, and one day following intervention (due to cross-over design, each subject underwent 4 total days of laboratory measurements). Field measurements were collected automatically at the participants' workstation in their working office.

Laboratory tests were conducted in a controlled, simulated work-space located at the University of Applied Sciences Campus Linz. All laboratory measurements were made in a controlled laboratory at the campus site Linz of the University of Applied Sciences Upper Austria. Temperature, air flow, humidity, lighting conditions (artificial light only) and noise level were controlled and set to be consistent with the subjects' typical working environment.

During the laboratory measurements, subjects either stood or sat upright in an ergonomic office chair, according to the study protocol. Subjects were encouraged to work as fast and as accurately as they could. To ensure identical testing conditions between subjects and to not unduly influence physiological parameters such as salivary cortisol level or heart rate variability, subjects were required to minimize excessive movement (e.g. standing up during the sitting periods).

In the first (initial) phase, participants were familiarized with the study protocol. Sitting time and weekly physical activity were determined via the IPAQ-questionnaire. Examples of each cognitive test implemented in the cognitive phase were executed according to their guidelines. A 30 minute break in a sitting posture was used to ascertain baseline heart-rate and cortisol level. Baseline heart-rate was calculated after a 20 minute rest for a 5 minute interval and saliva samples were collected at the end (30min) of the break.

In the second (cognitive) phase subjects participated in a test battery containing five blocks. Each block consisted of a working speed test (text editing task), an attentional test (d2R-test of attention) and a reaction time test (Stroop-test). These tests lasted for 30 minutes to fulfill recommendations regarding postural changes. To simulate "common" working conditions (computer based and non-computer based tasks), digital (text editing task, Stroop-test) as well as pen & paper (d2R-test) versions of the implemented tests were used. All blocks were executed in alternating postures (sit - stand - sit - stand - sit) and at the end of each block - after a 5 minute break - salivary samples were collected. The order of posture was not changed within groups or time.

In the third (final) phase participants were asked to estimate their workload by means of the NASA-TLX questionnaire followed by a 30 minute resting phase in a sitting posture. During both 30 min resting phases (initial & final) participants watched documentaries and were encouraged not to talk.

Salivary samples were collected after each break during the study protocol and on the following morning, 20 minutes after waking up, to ascertain cortisol awakening response (CAR). Salivary samples were centrifuged and stored at -80 °C for subsequent testing using a chemiluminescent immunoassay.

Heart-rate and trunk movements were measured from the start of the study protocol until the CAR measurement.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian (no acute or chronic diseases)
* Normal weight or slightly overweight (BMI: 18.5 - 27.5 kg/m²)
* Regularly working in sedentary office environments
* Regular computer users
* Fluent German speakers
* Consented to participate

Exclusion Criteria:

* Heavily overweight & Obesity (BMI > 27.5 kg/m²)
* Short office stay duration (< 8 h / day or < 20 h / week)
* Experience in sit-to-stand workstations
* Acute or chronic diseases
* Inability to stand
* Visual impairments that had not been corrected
* Color blindness
* People planning to change their physical activity level
* Regular smokers (> 1 cigarette /day)
* Not consented to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Daily sitting time | baseline and 23 weeks
  Changes in sitting time after 23 weeks in the experimental group compared with its own control period and the control group. Measuring methods: International Physical Activity Questionaire (IPAQ); self developed tracking software at the participants' workplace

SECONDARY OUTCOMES:
Cognitive performance (composite outcome) | baseline and 23 weeks
  Changes in cognitive performance after 23 weeks in the experimental group compared with its own control period and the control group. Measuring methods: Digital color-word-conflict stroop test, d2R-test of attention, text editing task, NASA-TLX

OTHER OUTCOMES:
Stress response | baseline and 23 weeks
  Changes in stress response after 23 weeks in the experimental group compared with its own control period and the control group. Measuring methods: Heart rate variability (HRV), salivary cortisol ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Schwartz, MSc, Study Director — University of Applied Sciences Upper Austria
Locations (1):
- University of Applied Sciences Upper Austria, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: Yes
Data resulting from this study will be analyzed and published in the PIs' PhD-thesis and journal articles.

REFERENCES:
- [Background] Neuhaus M, Healy GN, Dunstan DW, Owen N, Eakin EG. Workplace sitting and height-adjustable workstations: a randomized controlled trial. Am J Prev Med. 2014 Jan;46(1):30-40. doi: 10.1016/j.amepre.2013.09.009. PMID 24355669
- [Background] Commissaris DA, Konemann R, Hiemstra-van Mastrigt S, Burford EM, Botter J, Douwes M, Ellegast RP. Effects of a standing and three dynamic workstations on computer task performance and cognitive function tests. Appl Ergon. 2014 Nov;45(6):1570-8. doi: 10.1016/j.apergo.2014.05.003. Epub 2014 Jun 17. PMID 24951234
- [Background] Bates ME, Lemay EP Jr. The d2 Test of attention: construct validity and extensions in scoring techniques. J Int Neuropsychol Soc. 2004 May;10(3):392-400. doi: 10.1017/S135561770410307X. PMID 15147597
- [Background] Best JR, Nagamatsu LS, Liu-Ambrose T. Improvements to executive function during exercise training predict maintenance of physical activity over the following year. Front Hum Neurosci. 2014 May 27;8:353. doi: 10.3389/fnhum.2014.00353. eCollection 2014. PMID 24904387
- [Background] Hennig J, Friebe J, Ryl I, Kramer B, Bottcher J, Netter P. Upright posture influences salivary cortisol. Psychoneuroendocrinology. 2000 Jan;25(1):69-83. doi: 10.1016/s0306-4530(99)00037-2. PMID 10633536
- [Background] Van der Elst W, Van Boxtel MP, Van Breukelen GJ, Jolles J. The Stroop color-word test: influence of age, sex, and education; and normative data for a large sample across the adult age range. Assessment. 2006 Mar;13(1):62-79. doi: 10.1177/1073191105283427. PMID 16443719
- [Background] Lynch BM. Sedentary behavior and cancer: a systematic review of the literature and proposed biological mechanisms. Cancer Epidemiol Biomarkers Prev. 2010 Nov;19(11):2691-709. doi: 10.1158/1055-9965.EPI-10-0815. Epub 2010 Sep 10. PMID 20833969
- [Background] Owen N, Sparling PB, Healy GN, Dunstan DW, Matthews CE. Sedentary behavior: emerging evidence for a new health risk. Mayo Clin Proc. 2010 Dec;85(12):1138-41. doi: 10.4065/mcp.2010.0444. No abstract available. PMID 21123641
- [Background] Brown WJ, Miller YD, Miller R. Sitting time and work patterns as indicators of overweight and obesity in Australian adults. Int J Obes Relat Metab Disord. 2003 Nov;27(11):1340-6. doi: 10.1038/sj.ijo.0802426. PMID 14574344
- [Derived] Schwartz B, Kapellusch JM, Baca A, Wessner B. Medium-term effects of a two-desk sit/stand workstation on cognitive performance and workload for healthy people performing sedentary work: a secondary analysis of a randomised controlled trial. Ergonomics. 2019 Jun;62(6):794-810. doi: 10.1080/00140139.2019.1577497. Epub 2019 Apr 7. PMID 30762479
- [Derived] Schwartz B, Kapellusch JM, Schrempf A, Probst K, Haller M, Baca A. Effect of a novel two-desk sit-to-stand workplace (ACTIVE OFFICE) on sitting time, performance and physiological parameters: protocol for a randomized control trial. BMC Public Health. 2016 Jul 15;16:578. doi: 10.1186/s12889-016-3271-y. PMID 27422158